CLINICAL TRIAL: NCT00828152
Title: Internet-delivered Cognitive Behavioural Therapy for Health Anxiety - a Randomized Controlled Trial
Brief Title: Internet-delivered Cognitive Behavioral Therapy (CBT) for Health Anxiety
Acronym: Ha1b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Nils Lindefors, Psykiatri Sydväst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ha1b
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2010-06

CONDITIONS: Hypochondriasis
MeSH Terms: conditions — Hypochondriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Internet-delivered CBT. Contact with therapist thru an e-mail system. 12 weeks.
  Interventions: Behavioral: Internet-delivered CBT.
- 2 (Placebo Comparator): On line discussion group.
  Interventions: Behavioral: On line discussion group

INTERVENTIONS:
Behavioral: Internet-delivered CBT. — 12 weeks. Therapist contact through e-mail.
  Arms: 1
Behavioral: On line discussion group — Placebo. On line discussion group.
  Arms: 2

SUMMARY:
Hypochondriasis (health anxiety) is common, has many negative consequences for the afflicted individual and is associated with high societal costs. Cognitive Behavioural Therapy (CBT) has proven to be effective when administered in live-sessions. The aim of this study is to investigate whether CBT remains effective when administered via a self-help programme on the Internet.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of hypochondriasis
* At least 18 years old
* Able to read and write in swedish
* Computer access

Exclusion Criteria:

* Drug abuse
* Concurrent severe depression
* No serious somatic illness
* Previous treatment with CBT for hypochondriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Health Anxiety Inventory | 3 days before treatment start
Health Anxiety Inventory | 12 weeks after pre asessment
Health Anxiety Inventory | 6 months after post assessment
Health Anxiety Inventory | 12 months after post assessment

SECONDARY OUTCOMES:
IAS | Immediately pre and post treatment,and 6 and 12 month follow up
BAI | Immediately pre and post treatment, and 6 and 12 month follow-up
MADRS-S | Immediately pre and post treatment, and 6 and 12 month follow-up
QOLI | Immediately pre and post treatment, and 6 and 12 month follow-up
WI | Immediately pre and post treatment, and 6 and 12 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri Sydväst, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Hedman E, Andersson G, Lindefors N, Gustavsson P, Lekander M, Ruck C, Andersson E, Ljotsson B. Personality change following internet-based cognitive behavior therapy for severe health anxiety. PLoS One. 2014 Dec 1;9(12):e113871. doi: 10.1371/journal.pone.0113871. eCollection 2014. PMID 25437150
- [Derived] Hedman E, Andersson E, Lindefors N, Andersson G, Ruck C, Ljotsson B. Cost-effectiveness and long-term effectiveness of internet-based cognitive behaviour therapy for severe health anxiety. Psychol Med. 2013 Feb;43(2):363-74. doi: 10.1017/S0033291712001079. Epub 2012 May 21. PMID 22608115
- [Derived] Hedman E, Andersson G, Andersson E, Ljotsson B, Ruck C, Asmundson GJ, Lindefors N. Internet-based cognitive-behavioural therapy for severe health anxiety: randomised controlled trial. Br J Psychiatry. 2011 Mar;198(3):230-6. doi: 10.1192/bjp.bp.110.086843. PMID 21357882